CLINICAL TRIAL: NCT00386360
Title: A Non-Invasive Evaluation of Bone Microarchitecture Modification in Osteopenic Postmenopausal Women by 3D-Peripheral Quantitative Computed Tomography (3D-pQCT)
Brief Title: Study of the Effect of Once a Week Risedronate on the Microstructure of Tibia and Radius Using a New Scanning Method
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2005040
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-10

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo dose
  Interventions: Drug: Placebo comparator
- Risedronate (Experimental): 35 mg risedronate, orally, once weekly
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: Placebo comparator — oral weekly for one year
  Arms: Placebo
Drug: risedronate — 35 mg risedronate, once a week for one year
  Arms: Risedronate

SUMMARY:
The primary purpose of the protocol is to evaluate the sensitivity of 3D-pQCT (3D-Peripheral Quantitative Computed Tomography) technology to detect minute changes in bone microarchitecture.

DETAILED DESCRIPTION:
The 3D-pQCT equipment allows the evaluation of changes occurring within the bone at "microarchitecture" level, without the need for invasive bone biopsies. The primary objective is to evaluate the sensitivity of the technology to detect a difference between those treated with risedronate 35mg OAW (once a week) or placebo. Early phase postmenopausal women with osteopenia have been chosen because they have a more rapid and higher level of bone loss during the first few years of the menopause.

ELIGIBILITY:
Inclusion Criteria:

* cessation of menstruation (surgical or natural) between 6 and 36 months prior to study enrollment;
* osteopenic
* must have at least 1 evaluable radius and tibia, without history of fracture (traumatic or atraumatic)
* BMI (body mass index) between 18 and 28 kg/m2 inclusive;

Exclusion Criteria:

* history of any generalized bone disease, including hyperparathyroidism, Paget's disease of bone, renal osteodystrophy, or any other acquired or congenital bone disease; or any known condition that would interfere with the assessment of DXA (dual-energy X-ray absorptiometry) at either the lumbar spine (3 non-evaluable lumbar vertebrae at lumbar spine L1 - L4) or the femoral neck.
* clinical or radiological evidence of osteoporosis, such as atraumatic vertebral compression fracture (* 20% reduction in anterior-to-posterior or middle-to-posterior height ratio; or 20% reduction of the anterior, middle, and/or posterior height as compared with the adjacent vertebrae) documented by spinal X ray or a history of osteoporosis-related atraumatic fracture of the hip or of the wrist;
* glucocorticoid-induced osteopenia;
* previous bisphosphonate therapy;

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gioacchino D'Alo, MD, Principal Investigator — P&G Pharmaceuticals, Clinical Development Europe
Locations (9):
- Research Facility, Buenos Aires, Buenos Aires, Argentina
- Research Facility, Heidelberg, Victoria, Australia
- Research Facility, Toronto, Ontario, Canada
- France (3):
  - Research Facility, Lyon, Lyon
  - Research Facility, Saint-Etienne, Saint-Etienne
  - Research Facility, Toulouse, Toulouse
- Research Facility, Berlin, State of Berlin, Germany
- Research Facility, Geneva, Canton of Geneva, Switzerland
- Research Facility, Cambridge, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening started 3 April 2006
Groups:
- Placebo: Placebo, 1 tablet weekly on the same day
- Risedronate: 35 mg risedronate tablet, orally, once weekly on the same day
Period: Overall Study
Arm/Group | Placebo | Risedronate
Started | 49 | 112
Intent to Treat Population (ITT) | 49 (Includes all patients randomized and took at least one dose of study drug.) | 110
Primary Efficacy | 36 (Per-protocol patients with evaluable BVTV (trabecular bone volume/tissue volume) at baseline & M12.) | 77
Completed | 40 | 95
Not Completed | 9 | 17
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Did not take any study medication | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risedronate | Total
Number analyzed (Participants) | 49 | 112 | 161
Age Continuous [Mean (Standard Deviation); unit: years] — ITT Population
  years | 52.5 (2.2) | 52.6 (1.8) | 52.6 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 112 | 161
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — ITT Population
  Participants
    Asian (Oriental) | 1 | 0 | 1
    Caucasian | 48 | 107 | 155
    Hispanic | 0 | 2 | 2
    Multi-Racial | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  France | 9 | 24 | 33
  Germany | 23 | 46 | 69
  United Kingdom | 6 | 12 | 18
  Switzerland | 3 | 7 | 10
  Argentina | 6 | 15 | 21
  Australia | 0 | 2 | 2
  Canada | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Trabecular Bone Volume to Tissue Volume at Distal Radius, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: Primary Efficacy Population - all patients in ITT population who had no major protocol violations and had an evaluable distal radius BV/TV (trabecular bone volume to tissue volume) at baseline and Month 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 49 | 110
Percent Change | -1.486 [-2.577 to -0.396] | -1.255 [-2.012 to -0.498]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; In Laib 1998, the mean and SD of the annual loss in distal radius BV/TV were reported to be 3.5% and 6.4%, respectively. Assuming the treatment difference and SD of the percent change in distal radius BV/TV for this study were the same, it required enrolling 52 patients for placebo and 104 for risedronate to ensure 80% power to achieve 0.05 level of significance. Sample size estimation based on 2-sided 2-sample t-test and assumed effective size of 0.54 and dropout rate of 20%; Test type: Superiority or Other; p = 0.7096, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.231, 95% CI 2-sided [-0.995 to 1.458]

2. Secondary Outcome: Average Bone Density at Distal Radius, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: Per Protocol (PP) Population - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -2.121 [-3.028 to -1.214] | -1.578 [-2.208 to -0.947]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2973, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.543, 95% CI 2-sided [-0.485 to 1.571]

3. Secondary Outcome: Compact Bone Density at Distal Radius, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -0.786 [-1.337 to -0.234] | -0.301 [-0.685 to 0.082]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1275, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.485, 95% CI 2-sided [-0.141 to 1.110]

4. Secondary Outcome: Trabecular Bone Density at Distal Radius, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -1.820 [-3.020 to -0.619] | -1.156 [-1.991 to -0.321]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3360, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.664, 95% CI 2-sided [-0.697 to 2.025]

5. Secondary Outcome: Average Bone Density at Distal Tibia, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -0.440 [-1.221 to 0.340] | -0.106 [-0.652 to 0.439]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4565, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.334, 95% CI 2-sided [-0.551 to 1.219]

6. Secondary Outcome: Compact Bone Density at Distal Tibia, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -0.784 [-1.349 to -0.219] | -0.173 [-0.568 to 0.222]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0614, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.611, 95% CI 2-sided [-0.030 to 1.252]

7. Secondary Outcome: Trabecular Bone Density at Distal Tibia, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | 0.785 [-0.272 to 1.841] | 0.725 [-0.014 to 1.463]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9212, ANOVA; LS means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = -0.060, 95% CI 2-sided [-1.258 to 1.138]

8. Secondary Outcome: Lumbar Spine BMD, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -1.797 [-2.714 to -0.881] | 1.473 [0.839 to 2.106]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 3.270, 95% CI 2-sided [2.231 to 4.310]

9. Secondary Outcome: Total Proximal Femur BMD (Bone Mineral Density), Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -0.976 [-1.590 to -0.363] | 0.468 [0.043 to 0.892]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 1.444, 95% CI 2-sided [0.748 to 2.140]

10. Secondary Outcome: Femoral Neck BMD, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -1.422 [-2.250 to -0.595] | -0.014 [-0.586 to 0.558]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0036, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 1.408, 95% CI 2-sided [0.469 to 2.348]

11. Secondary Outcome: Greater Trochanter BMD, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -0.462 [-1.417 to 0.492] | 0.996 [0.336 to 1.656]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0087, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 1.458, 95% CI 2-sided [0.375 to 2.541]

12. Secondary Outcome: Type I Collagen C-Telopeptides, Serum, Percent Change From Baseline to Month 12
Description: ELISA / enzyme-linked immunosorbent assay method by central lab
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | 1.537 [-16.458 to 19.533] | -38.002 [-50.446 to -25.559]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = -39.540, 95% CI 2-sided [-59.957 to -19.123]

13. Secondary Outcome: Procollagen Type 1 N-Propeptide, Percent Change From Baseline to Month 12
Description: Electrochemiluminescence assay method by central lab
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -5.762 [-15.470 to 3.946] | -46.031 [-52.785 to -39.277]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = -40.269, 95% CI 2-sided [-51.300 to -29.238]

14. Secondary Outcome: Height, Percent Change From Baseline to Month 12
Time Frame: Baseline and Month 12
Population: PP - all patients in ITT population who had no major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo | Risedronate
Number analyzed (Participants) | 41 | 89
Percent Change | -0.163 [-0.270 to -0.056] | -0.071 [-0.146 to 0.003]
Statistical Analysis 1: Comparison: Placebo vs Risedronate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1385, ANOVA; LS Means are least squares (adjusted) means from ANOVA model with fixed effects for treatment and pooled center; LS Mean Difference = 0.092, 95% CI 2-sided [-0.030 to 0.213]

ADVERSE EVENTS:
Time Frame: Twelve Months
Arm/Group | Placebo | Risedronate
Serious Adverse Events (participants affected / at risk) | 5/49 | 7/110
Other Adverse Events (participants affected / at risk) | 38/49 | 76/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Risedronate (N=110)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skeletal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cholera (Infections and infestations) | 1 (1) | 0 (0)
Vestibuar Neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Cervical Root Pain (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Reaction (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary Bladder Polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Risedronate (N=110)
Nasopharyngitis (Infections and infestations) | 5 (5) | 10 (11)
Bronchitis (Infections and infestations) | 3 (3) | 7 (7)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4)
Influenza (Infections and infestations) | 4 (4) | 4 (4)
Cholera (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Vestibular Neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 4 (4)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (2)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Back Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 5 (5)
Hot Flush (Vascular disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Cervicobrachial Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Drug Intolerance (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Sensation of Foreign Body (General disorders) | 1 (1) | 0 (0)
Temperature Intolerance (General disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onchoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Weight Decreased (Investigations) | 1 (1) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less